CLINICAL TRIAL: NCT00165568
Title: Using Positron Emission Tomography to Evaluate the Effects of Bevacizumab on Intra-tumoral Pharmacokinetics of 5-fluorouracil in Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Massachusetts General Hospital (Other); Brigham and Women's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 04-415
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2009-11-02 (Estimated); Status verified 2009-10

CONDITIONS: Colorectal Cancer; Neoplasm Metastasis
Keywords: Positron emission tomography; PET; bevacizumab; 5fluorouracil; Metastatic colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis | interventions — Bevacizumab

INTERVENTIONS:
Drug: Bevacizumab

SUMMARY:
The purpose of this study is to investigate whether bevacizumab helps 5-Fluorouracil (5-FU) be delivered to the tumor more efficiently. Bevacizumab has been shown to inhibit the formation of new blood vessels in tumors and works best in combination with drugs that require blood vessels for transportation. Based on other experiments, bevacizumab may work by improving the transportation of other drugs to the tumor.

DETAILED DESCRIPTION:
* This is not a treatment study. A treatment regimen has already been decided upon by the patient and doctor.
* At the screening visit for this trial the following will be performed: a medical history, physical examination, CT scan to measure the amount and size of the tumor(s), and a PET scan using glucose that has been attached to a small amount of radioactivity to determine how well the tumor takes up glucose.
* Patients will then be randomized into one of 2 treatment groups. Group 1 will receive both 5-FU and bevacizumab on the first day of chemotherapy. Group 2 will receive just 5-FU on the first day of chemotherapy.
* Patients will undergo a PET scan that uses water that has been attached to a small amount of radioactivity to measure how well the tumor takes up water prior to the 5-FU adminstration.
* After patients receive 5-Fu they will undergo a PET scan during which a small amount of 5-FU has been attached to a small amount of radioactivity to measure how well the tumor takes up 5-FU.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic colorectal cancer subjects
* Subjects must have at least one non-radiated FDG-glucose avid (as demonstrated by an FDG-glucose PET scan) liver metastasis of at least 2 cm in size.
* Subjects must have never received chemotherapy for metastatic disease; subjects may have received adjuvant chemotherapy for presumed early stage disease if it was completed at least 12 months prior to study entry date
* All subjects must have already consented to an on-label use of a BV and fluorouracil containing first-line chemotherapy regimen (either with irinotecan or oxaliplatin) and must be a candidate for such a therapy as defined by the enrolling investigator and the community standard of care. As such a chemotherapy regimen requires an infusion port, this port should be placed at least two weeks prior to the subject's first dose of bevacizumab.
* Chronological age ≥ 18 years.
* ECOG performance status ≤ 2.
* Life expectancy ≥ 12 weeks.
* Women must not be pregnant or lactating. Both men and women of childbearing potential must be advised of the importance of using effective birth control measures during the course of the study.
* Subjects with concurrent malignancy of any site are eligible if the disease is under adequate control.
* All subjects must sign informed consent.

Exclusion Criteria:

* Subjects in "visceral crises", meaning a delay in achieving tumor response by 2 weeks may result in organ failure, are ineligible for this study.
* Subjects who are planned to undergo treatment with fluorouracil and bevacizumab alone (without irinotecan or oxaliplatin) are ineligible for this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2005-07; Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
To compare the percent change in tumor radioactivity uptake and retention after radiolabeled fluorouracil administration in subjects who receive bevacizumab versus those who do not receive bevacizumab.

SECONDARY OUTCOMES:
To compare the percent change in tumor flow induced by bevacizumab and fluorouracil
to evaluate the relationship between initial change in tumor radioactivity uptake and retention.

CONTACTS AND LOCATIONS:
Overall Officials: David Ryan, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts